CLINICAL TRIAL: NCT05630612
Title: Effects of Simultaneous ETA & AT1 Receptor Antagonism on Endothelial Function & Vascular Stiffness in ANCA-associated Vasculitis (SPARsentan in VASCulitis - SPARVASC)
Brief Title: ETA and AT1 Antagonism in ANCA-vasculitis (SPARVASC)
Acronym: SPARVASC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC22084
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: ANCA Associated Vasculitis; Cardiovascular Diseases; Kidney Diseases
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Cardiovascular Diseases; Kidney Diseases | interventions — sparsentan

STUDY DESIGN:
Intervention Model Description: Randomised, double blind, active control, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators will be blinded as will the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sparsentan (Experimental): 20 participants with ANCA-associated vasculitis in long-term disease remission.
  Participants will undergo a forearm blood flow study where forearm vasodilatation will be assessed in response to acetylcholine (7.5, 15 and 30ug/min) and sodium nitroprusside (1, 2 and 4ug/min). Participants will also receive bradykinin (100, 300 and 1000pmol/min) in order to assess tPA release to measure fibrinolytic capacity.
  Participants will also have 24h blood pressure assessed as well as measurements of arterial stiffness, systemic haemodynamics and measures of urinary protein.
  After these baseline measures have been obtained the subject will receive 6 weeks of sparsentan. Finally the subject will undergo the same investigations listed above and we will compare to see if measurements obtained differ after treatment.
  Interventions: Drug: Sparsentan
- Irbesartan (Active Comparator): 20 participants with ANCA-associated vasculitis in long-term disease remission.
  Participants will undergo a forearm blood flow study where forearm vasodilatation will be assessed in response to acetylcholine (7.5, 15 and 30ug/min) and sodium nitroprusside (1, 2 and 4ug/min). Participants will also receive bradykinin (100, 300 and 1000pmol/min) in order to assess tPA release to measure fibrinolytic capacity.
  Participants will also have 24h blood pressure assessed as well as measurements of arterial stiffness, systemic haemodynamics and measures of urinary protein.
  After these baseline measures have been obtained the subject will receive 6 weeks of irbesartan. Finally the subject will undergo the same investigations listed above and we will compare to see if measurements obtained differ after treatment.
  Interventions: Drug: Sparsentan

INTERVENTIONS:
Drug: Sparsentan — 6 weeks of treatment with sparsentan or irbesartan. This will be administered in a double-blind fashion.

SUMMARY:
ANCA-associated vasculitis is an autoimmune disease that causes damage to blood vessels. This leads to organ damage with the number of organs affected and the severity of damage varying significantly between patients.

Vasculitis patients also have a very high risk of heart attacks and strokes, called cardiovascular disease. A chemical called 'endothelin', produced by the blood vessels, causes vessels to stiffen and raises blood pressure and this associates with cardiovascular risk.

The investigators have previously shown that by blocking the effects of endothelin you reduce vessel stiffness, lower blood pressure and improve vessel function. However, these studies only blocked endothelin for a few hours. Now, the investigators would like to see if it is possible to maintain these benefits by blocking endothelin for longer.

Sparsentan is a tablet that blocks endothelin and lowers blood pressure. The investigators plan to give sparsentan to patients with vasculitis for 6 weeks. To determine if any beneficial effects of sparsentan are due to blood pressure lowering the investigators will give another group of vasculitis patients a tablet called irbesartan which lowers blood pressure but does not block endothelin. The investigators will compare the results between the two groups.

DETAILED DESCRIPTION:
ANCA-associated vasculitis is an autoimmune disease that causes direct damage to the vascular endothelium. Recent improvements in the immunosuppressive drugs used have improved short term outcomes but this has not translated to improved longer term outcomes. This is largely due to the significantly increased rates of cardiovascular disease experienced by this group of patients. For vasculitis patients in long-term remission the commonest cause of death is cardiovascular disease.

Autoimmune damage to the endothelium causes endothelial dysfunction and this associates with future risk of cardiovascular disease.

Endothelin-1 is a peptide produced by the endothelium. It is the most potent endogenous vasoconstrictor. It raises blood pressure, causes arterial stiffness and endothelial dysfunction, impairs fibrinolytic capacity and is pro-inflammatory.

Previous work has demonstrated that short term blockade of endothelin receptors improves vessel stiffness and fibrinolytic capacity.

The investigators will conduct a randomised, double blind, active control, parallel group study. 40 patients with ANCA-associated vasculitis in long-term remission will be recruited. 20 will be treated with 6 weeks of the endothelin-A receptor and angiotensin-1 receptor blocker sparsentan and 20 will be treated with the angiotensin-1 receptor blocker irbesartan.

Patients will undergo a forearm blood flow study before and after 6 weeks of treatment. This will assess endothelial function and allow the investigators to assess if the improvement in endothelial function noted with short term endothelin receptor blockade previously is maintained longer term.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* A diagnosis of ANCA-associated vasculitis that has been in remission for ≥6 months.

The diagnosis of AAV will have been made in accordance with the 2012 Revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides criteria. Remission will be defined as a Birmingham Vasculitis Activity Score (BVAS) of 0 for at least 2 months prior to the screening visit whilst taking prednisolone at daily dose ≤7.5mg, in conjunction with the treating clinician's assessment of clinically silent disease.

* eGFR ≥25ml/min/1.73m2 at screening.
* Women of childbearing potential, beginning at menarche, must agree to the use of one highly reliable method of contraception (ie, a failure rate of <1% per year) for at least 30 days prior to the first dose of the study medication (ie, for hormonal contraception) or according to manufacturer's recommendation (ie, for an intrauterine device) until 30 days after the last dose of the study medication, and must have a negative pregnancy test at screening. Women of childbearing potential are defined as those who are fertile, following menarche and until becoming postmenopausal, unless permanently sterile; permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as amenorrhea for more than 24 consecutive months without an alternative medical cause; women on hormone replacement therapy must have a documented plasma follicle-stimulating hormone level >40 mIU/mL.

Exclusion Criteria:

* Age <18 years
* Active vasculitis
* Liver disease
* Untreated hypertension (defined as systolic blood pressure >160 bpm and diastolic blood pressure >100 bpm)
* eGFR <25ml/min/1.73m2
* Any organ transplant recipients
* Haemodialysis/peritoneal dialysis patients
* A requirement for any medications contraindicated whilst taking sparsentan
* Congestive heart failure
* Patients not medically fit to attend for study visits
* Patients without mental capacity or willingness to provide informed consent
* History of multiple and/or severe (clinical judgement as determined by the investigator) allergic reactions to drugs, including the study drug or food.
* Patients who are pregnant or breast feeding, or those who plan to become pregnant during the study
* Participation in another clinical trial for 28 days before or 90 days after the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Forearm blood flow | Comparing baseline to after 6 weeks of intervention.
  Change from baseline to week 6 in acetylcholine-mediated forearm blood flow vasodilatation

SECONDARY OUTCOMES:
Fibrinolytic capacity | Comparing baseline to after 6 weeks of intervention.
  Plasma concentration of tissue plasminogen activator in response to bradykinin will be assessed before and after 6 weeks of intervention. Both tPA activity (in IU/ml) and tPA antigen (in ng/mL) will be assessed.
Blood pressure | Comparing baseline to after 3 and 6 weeks of treatment.
  Change from baseline 24h blood pressure and office blood pressure to after 3 and 6 weeks of treatment. We will assess systolic and diastolic blood pressure values as well as mean arterial pressure in mmHg.
Arterial stiffness | Comparing baseline to after 3 and 6 weeks of treatment.
  Change from baseline arterial stiffness to after 3 and 6 weeks of treatment. We will use a high fidelity micromanometer connected to a Sphygmocor device to measure pulse wave velocity in metres/second and augmentation index corrected for a heart rate of 75bpm measured in percentage.
Systemic haemodynamics | Comparing baseline to after 3 and 6 weeks of treatment.
  Change from baseline measures of systemic haemodynamics to after 3 and 6 weeks of treatment. We will use a BioZ diagnostics machine produced by CardioDynamics. This machine uses electrodes placed on the thorax and neck to automatically measure the following parameters of the heart beat cycle.
  Heart rate in beats/minute Stroke volume in mL/beat Stroke index in mL/beat/metre squared Cardiac output in L/min Cardiac Index in L/min/metre squared Systemic vascular resistance in dyne sec cm-5 Systemic vascular resistance index in dyne sec cm-5 metre squared Systolic time ratio index in sec-1 Thoracic fluid content in kiloohm-1
Proteinuria | Comparing baseline to after 3 and 6 weeks of treatment.
  Change from baseline measures of proteinuria to after 3 and 6 weeks of treatment.

OTHER OUTCOMES:
Optical Coherence Tomography (OCT) | Comparing baseline to after 3 and 6 weeks of treatment.
  Change from baseline OCT measures to after 3 and 6 weeks of treatment.
Fluorescence-activated cell sorting | Comparing baseline to after 6 weeks of treatment.
  Change from Baseline peripheral blood cells (balance of inflammatory and anti-inflammatory cells) analyzed using flow cytometry to after 6 weeks of treatment.
Endothelin-1 clearance | Comparing baseline to after 6 weeks of treatment.
  Change from Baseline peripheral blood monocytes ability to clear endothelin-1 using fluorescence-activated cell sorting (FACS) to after 6 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, Principal Investigator — University of Edinburgh
Locations (1):
- Centre for Cardiovascular Science, Queen's Medical Research Institute, 47 Little France Crescent, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data.

REFERENCES:
- [Background] Farrah TE, Melville V, Czopek A, Fok H, Bruce L, Mills NL, Bailey MA, Webb DJ, Dear JW, Dhaun N. Arterial stiffness, endothelial dysfunction and impaired fibrinolysis are pathogenic mechanisms contributing to cardiovascular risk in ANCA-associated vasculitis. Kidney Int. 2022 Nov;102(5):1115-1126. doi: 10.1016/j.kint.2022.07.026. Epub 2022 Aug 20. PMID 35998848